CLINICAL TRIAL: NCT02527044
Title: Impact of Preoperative FFR on Arterial Bypass Graft Functionality: Towards a New CABG Paradigm
Brief Title: Impact of Preoperative FFR on Arterial Bypass Graft Functionality
Acronym: IMPAG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 4385
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Heart Disease
Keywords: Coronary Artery Bypass; Flow Reserve
MeSH Terms: conditions — Heart Diseases | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: FFR values are collected by a member of the research staff. The treating physicians, the patient, and the outcome assessor will be blinded to the pre-operative FFR values.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional graft (Experimental): Follow-up angiography of all bypass grafts and anastomoses six months after surgery: anastomotic function was scored as 0 for an occluded graft, 1 when the flow from the native coronary artery was dominant, 2 when flow supply from the native coronary and from the graft was balanced, and 3 when the native coronary was fully opacified by the graft. An anastomosis was considered "functional" for score of 3.
  Interventions: Procedure: Fractional Flow Reserve (FFR)
- Non functional graft (Active Comparator): Follow-up angiography of all bypass grafts and anastomoses six months after surgery: anastomotic function was scored as 0 for an occluded graft, 1 when the flow from the native coronary artery was dominant, 2 when flow supply from the native coronary and from the graft was balanced, and 3 when the native coronary was fully opacified by the graft. An anastomosis was considered "non functional" for scores of 0 to 2.
  Interventions: Procedure: Fractional Flow Reserve (FFR)

INTERVENTIONS:
Procedure: Fractional Flow Reserve (FFR) — An FFR will be performed pre-operative to the CABG procedure

SUMMARY:
This study was designed to evaluate the correlation between pre-operative FFR and the functionality of arterial bypass grafts six months after coronary artery bypass grafting. Patients with multi-vessel coronary artery disease will undergo both a coronary angiogram and FFR during their diagnostic workup. All patients will be referred for surgical revascularization (CABG) with planned use of arterial grafts. Six months after surgery, patients will undergo an angiogram to assess the functionality of the bypass graft and anastomosis.

DETAILED DESCRIPTION:
The objective of surgical coronary revascularization is to restore blood flow supply to a myocardial territory that is ischemic or at risk of infarction, by interposing a low-resistance conduit in parallel to a major diseased coronary artery segment. The conductance of this additional conduit must be sufficient to accommodate high flow demands with minimal pressure drop at the site of distal implantation. Such a conduit may be used either as single independent graft, or assembled in a variety of sequential configurations, according to the preferred technique and based on the underlying coronary artery disease (CAD). Saphenous vein grafts (SVGs), most commonly used as single free grafts reimplanted on the aorta, are large conduits with very limited vasomotion. Their resistance to blood flow is negligible due to their large diameter, absence of muscular layer and usually short length, but their long-term patency is hindered by the development of premature atherosclerosis. In contrast, arterial grafts are usually of smaller diameter and more resistive due to their histological features. These arterial conduits are usually used in situ, as the second or third order of branches from the aorta and, therefore, have higher pressure drops compared to grafts implanted directly onto the aorta. Alternatively, the creation of composite T grafts with the free right internal thoracic artery (RITA) connected to the in situ left internal thoracic artery (LITA) can allow revascularization of all myocardium at risk. However, consequences of such a combination are that the flow supply is entirely dependent on the flow capacity of the proximal LITA, and that resistance along the graft may become a concern, particularly at the more distal anastomoses of the configuration (due to the cumulative length and distal graft tapering).

Competitive flow typically occurs when the resistance of the graft closely matches that of the native coronary artery target. In this situation, both the native coronary artery and the bypass graft contribute to distal perfusion, each providing resistance to blood flow from the other. Schematically, these resistances are arranged in parallel with input pressure at the coronary ostium or at the ostium of the graft, and output pressure at the anastomotic target site. The pressures at the two ends of the circuit are identical with only minor phasic variations in proximal pressure due to the delay in progression of the systolic pressure wave from the coronary ostium to the more distal ostium of the graft. According to Ohm's law, blood flow is directly proportional to pressure gradient and inversely proportional to resistance. Consequently, the relative contribution of the graft and of the native circulation to distal perfusion will be inversely proportional to their own resistance: if the resistance of the graft exceeds that of the native vessel (for instance, in situations of non-severely obstructive CAD), the distal territory will be predominantly perfused by the native coronary artery; if the resistance of the native vessel remains higher, the flow through the graft will be predominant; if both conduits oppose near-identical resistances to flow, their contribution to distal blood flow will be equivalent.

Many reports have consistently suggested that competitive flow in arterial bypass grafts negatively affects patency: more graft failures are observed when native coronary stenosis is less severe. Further, the misunderstanding of competitive flow also impairs multiple arterial grafting adoption rates, which remain quite low worldwide despite proven superior outcomes, due in large part to incomplete understanding of the effects of flow competition by surgeons. Current methods to evaluate coronary stenosis are: visual inspection, quantitative computerized angiography (QCA) and fractional flow reserve (FFR). Several studies have compared these three methods, demonstrating that visual assessment and QCA are of limited value for accurately predicting the significance of most intermediate narrowings and, therefore, at predicting a competition phenomenon. In contrast, FFR measures the consequence of the stenosis in terms of reduction of blood flow capacity. FFR reliably identifies stenoses associated with inducible ischemia with more than 93% accuracy, a rate higher than any other test. Despite these advantages, FFR is not widely applied especially in coronary surgery whereas in interventional cardiology, it is used near systematically. What the investigators propose in this collaborative study is a complete paradigm shift in how coronary surgery is carried out - total arterial grafting supported by a true physiologic basis, and a correlated proof of its outcomes.

Currently, indications for surgical coronary revascularization still largely rely only on visual estimation of stenoses. Unfortunately, the estimation of the true coronary lesion severity by visual estimation is especially poor for moderate lesions, i.e. between 50 to 70% stenosis. An FFR cutoff value of 0.8 is obtained in only 35% of these moderate lesions. When using saphenous vein, the impact of competition flow on graft patency is minimal in this situation but when an artery conduit is preferred, it impacts the functionality of the graft significantly.

Therefore, the investigators are proposing a prospective FFR evaluation of surgical patients with 3-vessel CAD, whose disease severity will be estimated by visual inspection during diagnostic angiogram. FFR will be performed and all values will be recorded; however, the patient, interventional cardiologist, and surgeon will be blinded to its results. All patients will then undergo coronary surgery with planned arterial revascularization. Six months after surgery, a control angiogram will be performed to evaluate functionality of the grafts. The results of this functional assessment will be correlated with the preoperative FFR values, in order to find a cutoff above which the arterial grafts are not functional, which will also be analyzed by subgroups defined according to configuration (i.e. in situ or composite).

ELIGIBILITY:
Inclusion Criteria:

1. All patients with multi-vessel coronary artery disease undergoing elective or urgent first time coronary artery bypass grafting (CABG).
2. All patients undergoing diagnostic angiography and suspected to have multi-vessel disease for referral to CABG
3. Patients requiring both on-pump or off-pump CABG are accepted, as long as a arterial revascularisation is planned.
4. The patients must be over the age of 18.
5. CABG is the only procedure being conducted

Exclusion Criteria:

1. Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stenting)
2. Redo CABG, or a percutaneous coronary intervention (PCI) within the last 6 months.
3. Severe renal insufficiency (preoperative creatinine >150umol/L) contraindicating postoperative coronary angiography
4. Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
5. Women who are pregnant or are seeking to become pregnant
6. Must not have severe congestive heart failure (class III or IV New York Heart Association) at enrollment
7. Left ventricular ejection fraction less than 30%
8. Prior history of significant bleeding that might be expected to recur with CABG
9. Prisoners or institutionalized individuals
10. Geographic inaccessibility for the follow-up visits required by protocol
11. Concurrent enrollment in another clinical trial
12. Extra-cardiac illness that is expected to limit survival to less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Correlation between pre-operative FFR and anastomosis function | Up to 12 months
  The primary outcome was the evaluation of the correlation between target vessel pre-operative FFR value and the anastomosis function as measured by angiogram approximately 6 months after surgery.

SECONDARY OUTCOMES:
Correlation between pre-operative FFR and anastomosis occlusion | Up to 12 months
  The evaluation of the correlation between target vessel pre-operative FFR value and occlusion of the anastomosis measured by angiogram approximately 6 months after surgery.
Major Adverse Cardiac Events | Up to 12 months
  Major adverse cardiac events (MACE) is a qualitative measurement of any adverse cardiac events such as death or myocardial infraction after the operative procedure.

CONTACTS AND LOCATIONS:
Overall Officials: David Glineur, MD, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Clinique Saint-Luc Bouge, Bouge, Belgium
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glineur D, Poncelet A, El Khoury G, D'hoore W, Astarci P, Zech F, Noirhomme P, Hanet C. Fractional flow reserve of pedicled internal thoracic artery and saphenous vein grafts 6 months after bypass surgery. Eur J Cardiothorac Surg. 2007 Mar;31(3):376-81. doi: 10.1016/j.ejcts.2006.11.023. Epub 2006 Dec 14. PMID 17174100
- [Background] Glineur D, Djaoudi S, D'horre W, Gurne O, Delouvroy A, de Kerchove L, El Khoury G, Hanet C. Endothelium-dependent and endothelium-independent vasodilator response of left and right internal mammary and internal thoracic arteries used as a composite Y-graft. Eur J Cardiothorac Surg. 2011 Aug;40(2):389-93. doi: 10.1016/j.ejcts.2010.11.055. Epub 2011 Jan 28. PMID 21277219
- [Background] Glineur D, Hanet C, Poncelet A, D'hoore W, Funken JC, Rubay J, Kefer J, Astarci P, Lacroix V, Verhelst R, Etienne PY, Noirhomme P, El Khoury G. Comparison of bilateral internal thoracic artery revascularization using in situ or Y graft configurations: a prospective randomized clinical, functional, and angiographic midterm evaluation. Circulation. 2008 Sep 30;118(14 Suppl):S216-21. doi: 10.1161/CIRCULATIONAHA.107.751933. PMID 18824757
- [Background] Glineur D, Noirhomme P, Reisch J, El Khoury G, Astarci P, Hanet C. Resistance to flow of arterial Y-grafts 6 months after coronary artery bypass surgery. Circulation. 2005 Aug 30;112(9 Suppl):I281-5. doi: 10.1161/CIRCULATIONAHA.104.524702. PMID 16159832
- [Background] Lemma M, Innorta A, Pettinari M, Mangini A, Gelpi G, Piccaluga M, Danna P, Antona C. Flow dynamics and wall shear stress in the left internal thoracic artery: composite arterial graft versus single graft. Eur J Cardiothorac Surg. 2006 Apr;29(4):473-8. doi: 10.1016/j.ejcts.2006.01.035. Epub 2006 Mar 7. PMID 16522367
- [Background] Glineur D, Hanet C. Competitive flow in coronary bypass surgery: is it a problem? Curr Opin Cardiol. 2012 Nov;27(6):620-8. doi: 10.1097/HCO.0b013e3283583000. PMID 23075821
- [Background] Glineur D, Hanet C. Competitive flow and arterial graft a word of caution. Eur J Cardiothorac Surg. 2012 Apr;41(4):768-9. doi: 10.1093/ejcts/ezr064. Epub 2011 Nov 24. No abstract available. PMID 22423057
- [Background] Glineur D, D'hoore W, de Kerchove L, Noirhomme P, Price J, Hanet C, El Khoury G. Angiographic predictors of 3-year patency of bypass grafts implanted on the right coronary artery system: a prospective randomized comparison of gastroepiploic artery, saphenous vein, and right internal thoracic artery grafts. J Thorac Cardiovasc Surg. 2011 Nov;142(5):980-8. doi: 10.1016/j.jtcvs.2011.07.017. PMID 22014339
- [Background] Glineur D, D'hoore W, El Khoury G, Sondji S, Kalscheuer G, Funken JC, Rubay J, Poncelet A, Astarci P, Verhelst R, Noirhomme P, Hanet C. Angiographic predictors of 6-month patency of bypass grafts implanted to the right coronary artery a prospective randomized comparison of gastroepiploic artery and saphenous vein grafts. J Am Coll Cardiol. 2008 Jan 15;51(2):120-5. doi: 10.1016/j.jacc.2007.09.030. PMID 18191734
- [Background] Glineur D, Hanet C, D'hoore W, Poncelet A, De Kerchove L, Etienne PY, Noirhomme P, El Khoury G. Causes of non-functioning right internal mammary used in a Y-graft configuration: insight from a 6-month systematic angiographic trial. Eur J Cardiothorac Surg. 2009 Jul;36(1):129-35; discussion 135-6. doi: 10.1016/j.ejcts.2009.02.041. Epub 2009 Apr 15. PMID 19372044
- [Background] Sabik JF 3rd, Lytle BW, Blackstone EH, Khan M, Houghtaling PL, Cosgrove DM. Does competitive flow reduce internal thoracic artery graft patency? Ann Thorac Surg. 2003 Nov;76(5):1490-6; discussion 1497. doi: 10.1016/s0003-4975(03)01022-1. PMID 14602274
- [Background] White CW, Wright CB, Doty DB, Hiratza LF, Eastham CL, Harrison DG, Marcus ML. Does visual interpretation of the coronary arteriogram predict the physiologic importance of a coronary stenosis? N Engl J Med. 1984 Mar 29;310(13):819-24. doi: 10.1056/NEJM198403293101304. PMID 6700670
- [Background] Bursch JH, Hahne HJ, Brennecke R, Gronemeier D, Heintzen PH. Assessment of arterial blood flow measurements by digital angiography. Radiology. 1981 Oct;141(1):39-47. doi: 10.1148/radiology.141.1.7291540.
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Nam CW, Mangiacapra F, Entjes R, Chung IS, Sels JW, Tonino PA, De Bruyne B, Pijls NH, Fearon WF; FAME Study Investigators. Functional SYNTAX score for risk assessment in multivessel coronary artery disease. J Am Coll Cardiol. 2011 Sep 13;58(12):1211-8. doi: 10.1016/j.jacc.2011.06.020. PMID 21903052
- [Background] Tonino PA, Fearon WF, De Bruyne B, Oldroyd KG, Leesar MA, Ver Lee PN, Maccarthy PA, Van't Veer M, Pijls NH. Angiographic versus functional severity of coronary artery stenoses in the FAME study fractional flow reserve versus angiography in multivessel evaluation. J Am Coll Cardiol. 2010 Jun 22;55(25):2816-21. doi: 10.1016/j.jacc.2009.11.096. PMID 20579537
- [Background] Christou MA, Siontis GC, Katritsis DG, Ioannidis JP. Meta-analysis of fractional flow reserve versus quantitative coronary angiography and noninvasive imaging for evaluation of myocardial ischemia. Am J Cardiol. 2007 Feb 15;99(4):450-6. doi: 10.1016/j.amjcard.2006.09.092. Epub 2006 Dec 20. PMID 17293182
- [Background] Meijboom WB, Van Mieghem CA, van Pelt N, Weustink A, Pugliese F, Mollet NR, Boersma E, Regar E, van Geuns RJ, de Jaegere PJ, Serruys PW, Krestin GP, de Feyter PJ. Comprehensive assessment of coronary artery stenoses: computed tomography coronary angiography versus conventional coronary angiography and correlation with fractional flow reserve in patients with stable angina. J Am Coll Cardiol. 2008 Aug 19;52(8):636-43. doi: 10.1016/j.jacc.2008.05.024. PMID 18702967
- [Background] Pijls NH, De Bruyne B, Peels K, Van Der Voort PH, Bonnier HJ, Bartunek J Koolen JJ, Koolen JJ. Measurement of fractional flow reserve to assess the functional severity of coronary-artery stenoses. N Engl J Med. 1996 Jun 27;334(26):1703-8. doi: 10.1056/NEJM199606273342604. PMID 8637515
- [Background] Botman CJ, Schonberger J, Koolen S, Penn O, Botman H, Dib N, Eeckhout E, Pijls N. Does stenosis severity of native vessels influence bypass graft patency? A prospective fractional flow reserve-guided study. Ann Thorac Surg. 2007 Jun;83(6):2093-7. doi: 10.1016/j.athoracsur.2007.01.027. PMID 17532405
- [Background] Mohr FW, Morice MC, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR Jr, Morel MA, Van Dyck N, Houle VM, Dawkins KD, Serruys PW. Coronary artery bypass graft surgery versus percutaneous coronary intervention in patients with three-vessel disease and left main coronary disease: 5-year follow-up of the randomised, clinical SYNTAX trial. Lancet. 2013 Feb 23;381(9867):629-38. doi: 10.1016/S0140-6736(13)60141-5. PMID 23439102
- [Background] Eagle KA, Guyton RA, Davidoff R, Edwards FH, Ewy GA, Gardner TJ, Hart JC, Herrmann HC, Hillis LD, Hutter AM Jr, Lytle BW, Marlow RA, Nugent WC, Orszulak TA; American College of Cardiology; American Heart Association. ACC/AHA 2004 guideline update for coronary artery bypass graft surgery: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1999 Guidelines for Coronary Artery Bypass Graft Surgery). Circulation. 2004 Oct 5;110(14):e340-437. No abstract available. PMID 15466654
- [Background] Smith SC Jr, Allen J, Blair SN, Bonow RO, Brass LM, Fonarow GC, Grundy SM, Hiratzka L, Jones D, Krumholz HM, Mosca L, Pasternak RC, Pearson T, Pfeffer MA, Taubert KA; AHA/ACC; National Heart, Lung, and Blood Institute. AHA/ACC guidelines for secondary prevention for patients with coronary and other atherosclerotic vascular disease: 2006 update: endorsed by the National Heart, Lung, and Blood Institute. Circulation. 2006 May 16;113(19):2363-72. doi: 10.1161/CIRCULATIONAHA.106.174516. No abstract available. PMID 16702489
- [Background] Hanet C, Robert A, Wijns W. Vasomotor response to ergometrine and nitrates of saphenous vein grafts, internal mammary artery grafts, and grafted coronary arteries late after bypass surgery. Circulation. 1992 Nov;86(5 Suppl):II210-6. PMID 1424002
- [Background] Kulik A, Le May M, Wells GA, Mesana TG, Ruel M. The clopidogrel after surgery for coronary artery disease (CASCADE) randomized controlled trial: clopidogrel and aspirin versus aspirin alone after coronary bypass surgery [NCT00228423]. Curr Control Trials Cardiovasc Med. 2005 Oct 11;6(1):15. doi: 10.1186/1468-6708-6-15. PMID 16219100
- [Background] Kulik A, Le May MR, Voisine P, Tardif JC, Delarochelliere R, Naidoo S, Wells GA, Mesana TG, Ruel M. Aspirin plus clopidogrel versus aspirin alone after coronary artery bypass grafting: the clopidogrel after surgery for coronary artery disease (CASCADE) Trial. Circulation. 2010 Dec 21;122(25):2680-7. doi: 10.1161/CIRCULATIONAHA.110.978007. Epub 2010 Dec 6. PMID 21135365
- [Background] Une D, Kulik A, Voisine P, Le May M, Ruel M. Correlates of saphenous vein graft hyperplasia and occlusion 1 year after coronary artery bypass grafting: analysis from the CASCADE randomized trial. Circulation. 2013 Sep 10;128(11 Suppl 1):S213-8. doi: 10.1161/CIRCULATIONAHA.112.000328. PMID 24030409
- [Background] Une D, Al-Atassi T, Kulik A, Voisine P, Le May M, Ruel M. Impact of clopidogrel plus aspirin versus aspirin alone on the progression of native coronary artery disease after bypass surgery: analysis from the Clopidogrel After Surgery for Coronary Artery DiseasE (CASCADE) randomized trial. Circulation. 2014 Sep 9;130(11 Suppl 1):S12-8. doi: 10.1161/CIRCULATIONAHA.113.008227. PMID 25200049
- [Background] Kulik A, Ruel M, Jneid H, Ferguson TB, Hiratzka LF, Ikonomidis JS, Lopez-Jimenez F, McNallan SM, Patel M, Roger VL, Sellke FW, Sica DA, Zimmerman L; American Heart Association Council on Cardiovascular Surgery and Anesthesia. Secondary prevention after coronary artery bypass graft surgery: a scientific statement from the American Heart Association. Circulation. 2015 Mar 10;131(10):927-64. doi: 10.1161/CIR.0000000000000182. Epub 2015 Feb 9. No abstract available. PMID 25679302
- [Derived] Glineur D, Grau JB, Etienne PY, Benedetto U, Fortier JH, Papadatos S, Laruelle C, Pieters D, El Khoury E, Blouard P, Timmermans P, Ruel M, Chong AY, So D, Chan V, Rubens F, Gaudino MF. Impact of preoperative fractional flow reserve on arterial bypass graft anastomotic function: the IMPAG trial. Eur Heart J. 2019 Aug 1;40(29):2421-2428. doi: 10.1093/eurheartj/ehz329. PMID 31155673